CLINICAL TRIAL: NCT07215767
Title: Clinical Study to Investigate the Antihypersensitivity Efficacy of a Novel Dentifrice
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300140
Record Dates: First submitted 2025-10-06; First posted 2025-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test Dentifrice (Experimental): Participants will be instructed to dose the toothbrush head with the Test Dentifrice (at least a 1-inch strip of product), then brush the teeth thoroughly for at least 1-minute, twice a day (morning and evening) for approximately 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Stannous fluoride and Potassium nitrate Dentifrice
- Reference Dentifrice 1 (Active Comparator): Participants will be instructed to dose the toothbrush head with Reference Dentifrice 1 (at least a 1-inch strip of product), then brush the teeth thoroughly for at least 1-minute, twice a day (morning and evening) for approximately 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Stannous fluoride Dentifrice
- Reference Dentifrice 2 (Active Comparator): Participants will be instructed to dose the toothbrush head with Reference Dentifrice 2 (at least a 1-inch strip of product), then brush the teeth thoroughly for at least 1-minute, twice a day (morning and evening) for approximately 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Potassium nitrate Dentifrice
- Reference Dentifrice 3 (Placebo Comparator): Participants will be instructed to dose the toothbrush head with Reference Dentifrice 3 (at least a 1-inch strip of product), then brush the teeth thoroughly for at least 1-minute, twice a day (morning and evening) for approximately 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Vehicle Dentifrice

INTERVENTIONS:
Drug: Stannous fluoride and Potassium nitrate Dentifrice — Fluoride dentifrice
  Arms: Test Dentifrice
Drug: Stannous fluoride Dentifrice — Fluoride dentifrice
  Arms: Reference Dentifrice 1
Drug: Potassium nitrate Dentifrice — Non-fluoride dentifrice
  Arms: Reference Dentifrice 2
Drug: Vehicle Dentifrice — Placebo dentifrice
  Arms: Reference Dentifrice 3

SUMMARY:
The aim of this clinical study is to demonstrate the superior antihypersensitivity efficacy of a novel stannous fluoride (SnF2) and potassium nitrate (KNO3) dentifrice (Investigational Product), compared to SnF2 only, KNO3 only and Vehicle dentifrices, after 8 weeks twice daily use.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, controlled, double-blind, 4-treatment arm, stratified, parallel design, Phase III clinical study in healthy participants, aged 12-65 years inclusive, with self-reported and clinically confirmed dentin hypersensitivity. Participants who meet the required study criteria at Screening and Baseline will be stratified and randomized to one of four study dentifrices. Approximately 630 qualifying participants will be randomized to study treatment (approximately 180 participants each to the SnF2 and KNO3 dentifrice, the SnF2 dentifrice and the KNO3 dentifrice; approximately 90 participants to the Vehicle dentifrice). Dentin hypersensitivity will be clinically assessed at Screening and Baseline, and after 3 days, 1 week, 2 weeks, 4 weeks and 8 weeks treatment (7 study visits).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent document (and assent document, if appropriate)
* Participant is biologically male or female.
* Participant is 12 to 65 years of age, inclusive, at the time of signing the consent/assent form.
* Participant is in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in self-reported medical history, or upon oral examination, that would impact their safety or well-being, or the outcomes of the study, if they were to participate in the study, or affect their ability to understand and follow study requirements.
* Participant has a history of tooth sensitivity lasting more than six months but not more than 10 years (self-reported).
* Participant has a minimum of 2 non-adjacent teeth (incisors, canines or premolars), in different quadrants, with exposed dentin due to facial/cervical erosion, abrasion or gingival recession, and clinically confirmed dentin hypersensitivity to tactile and evaporative (air) stimuli at Screening and Baseline.

Exclusion Criteria:

* Female participant who is pregnant at Screening and Baseline, or is intending to become pregnant during the study.
* Female participant who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to any of the study products, any of their stated ingredients or closely related compounds.
* Participant is participating in, or has participated in, other studies (including non-medicinal studies) involving an Investigational Product within 30 days of Screening or plans to participate in other studies (including non-medicinal studies) during this study.
* Participant has participated in a tooth sensitivity study within 8 weeks of Screening.
* Participant is currently using an oral care product indicated for dentin hypersensitivity relief or care of sensitive teeth or has used an antihypersensitivity oral care product within 8 weeks of Screening.
* Participant takes daily doses of medications/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity.
* Participant has had professional tooth de-sensitising treatment within 8 weeks of Screening.
* Participant has had a tooth bleaching procedure within 8 weeks of Screening.
* Participant has had dental prophylaxis within 4 weeks of Screening.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with evidence of current/recent active dental caries or treatment for decay within 12 months of Screening.
* Participant who, in the opinion of the investigator or dentally qualified designee, is at high risk of dental caries.
* Participant with specific dentition exclusions for 'Test Teeth'.
* Participant has taken antibiotics in the 2 weeks prior to Screening or Baseline.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Schiff sensitivity score at Week 8 (Test Dentifrice Versus [Vs] Reference Dentifrices 1, 2 and 3) | Baseline and Week 8
  Evaporative (air) sensitivity will be assessed by the participant's response to an evaporative (air) stimulus administered by the clinical examiner. Participant response will be evaluated immediately following application of the stimulus using the Schiff sensitivity scale (0=Participant does not respond to air stimulation, 1=Participant responds to air stimulus but does not request discontinuation of stimulus, 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3=Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of stimulus). A decrease in Schiff sensitivity score indicates improvement. Schiff sensitivity score = mean score of the two 'Test Teeth' (selected at Baseline). Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline = Week 8 score minus Baseline score.
Change from Baseline in tactile threshold (grams [g]) at Week 8 (Test Dentifrice Vs Reference Dentifrices 1, 2 and 3) | Baseline and Week 8
  Tactile sensitivity will be assessed by the participant's response to a tactile stimulus administered by the clinical examiner using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold in g. At Baseline, upper force setting will be 20g; at Week 8, upper force setting will be 80g. An increase in tactile threshold (g) indicates improvement. Tactile threshold (g) = mean value for the two 'Test Teeth'. Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline in tactile threshold (g) at Week 8 = Week 8 value minus Baseline value.

SECONDARY OUTCOMES:
Change from Baseline in Schiff sensitivity score at Day 4, Week 1, Week 2 and Week 4 (Test Dentifrice Vs Reference Dentifrices 1, 2 and 3) | Baseline, Day 4, Week 1, Week 2 and Week 4
  Evaporative (air) sensitivity will be assessed by the participant's response to an evaporative (air) stimulus administered by the clinical examiner. Participant response will be evaluated immediately following application of the stimulus using the Schiff sensitivity scale (0=Participant does not respond to air stimulation, 1=Participant responds to air stimulus but does not request discontinuation of stimulus, 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3=Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus). A decrease in Schiff sensitivity score indicates improvement. Schiff sensitivity score = mean score of the two 'Test Teeth'. Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline = score at given timepoint minus Baseline score.
Change from Baseline in tactile threshold (g) at Day 4, Week 1, Week 2 and Week 4 (Test Dentifrice Vs Reference Dentifrices 1, 2 and 3) | Baseline, Day 4, Week 1, Week 2 and Week 4
  Tactile sensitivity will be assessed by the participant's response to a tactile stimulus administered by the clinical examiner using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold in g. At Baseline, upper force setting will be 20g; at other timepoints, upper force setting will be 80g. An increase in tactile threshold (g) indicates improvement. Tactile threshold (g) = mean value for the two 'Test Teeth'. Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline in tactile threshold (g) = value at given timepoint minus Baseline value.
Change from Baseline in Schiff sensitivity score at Day 4, Week 1, Week 2, Week 4 and Week 8 (Reference Dentifrices 1 and 2 Vs Reference Dentifrice 3) | Baseline, Day 4, Week 1, Week 2, Week 4 and Week 8
  Evaporative (air) sensitivity will be assessed by the participant's response to an evaporative (air) stimulus administered by the clinical examiner. Participant response will be evaluated immediately following application of the stimulus using the Schiff sensitivity scale (0=Participant does not respond to air stimulation, 1=Participant responds to air stimulus but does not request discontinuation of stimulus, 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3=Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus). A decrease in Schiff sensitivity score indicates improvement. Schiff sensitivity score = mean score of the two 'Test Teeth'. Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline = score at given timepoint minus Baseline score.
Change from Baseline in tactile threshold (g) at Day 4, Week 1, Week 2, Week 4 and Week 8 (Reference Dentifrices 1 and 2 Vs Reference Dentifrice 3) | Baseline, Day 4, Week 1, Week 2, Week 4 and Week 8
  Tactile sensitivity will be assessed by the participant's response to a tactile stimulus administered by the clinical examiner using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold in g. At Baseline, the upper force setting will be 20g; at other timepoints, the upper force setting will be 80g. An increase in tactile threshold (g) indicates improvement. Tactile threshold (g) = mean value for the two 'Test Teeth'. Change from Baseline is calculated for each 'Test Tooth' first before calculating mean change for the two 'Test Teeth', where change from Baseline in tactile threshold (g) = value at given timepoint minus Baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Pejmon Amini, Principal Investigator — Silverstone Research; Jeffery L Milleman, Principal Investigator — Salus Research, Inc; John T Gallob, Principal Investigator — All Sum Research
Locations (3):
- United States (3):
  - All Sum Research Limited, Melbourne, Florida
  - Salus Research, Inc., Fort Wayne, Indiana
  - Silverstone Research, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary and key secondary endpoints and the safety data for the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.